CLINICAL TRIAL: NCT05193604
Title: Phase I Clinical Trial to Evaluate the Tolerability and Safety of TQB2858 Injection in Subjects With Metastatic Pancreatic Cancer
Brief Title: A Clinical Trial to Evaluate Tolerability and Security of TQB2858 Injection in Subjects With Advanced Pancreatic Carcinoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to the adjustment of sponsor's development strategies and pipeline.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Nanjing Shunxin Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQB2858-I-02
Record Dates: First submitted 2021-12-28; First posted 2022-01-18 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-01

CONDITIONS: Pancreatic Carcinoma
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; Injections; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQB2858 injection (Experimental): Cohort 1: TQB2858 injection administered intravenously on day 1 of each 21-day cycle.
  Cohort 2: TQB2858 injection administered intravenously on day 1 of each 21-day cycle, gemcitabine and albumin paclitaxel administered intravenously on day 1 and day 7 of each 21-day cycle.
  Cohort 3: TQB2858 injection administered intravenously on day 1 of each 21-day cycle，gemcitabine and albumin paclitaxel administered intravenously on day 1 and day 7 of each 21-day cycle，Anlotinib capsules 8 mg given orally, once daily in 21-day cycle (14 days on treatment from Day 1-14, 7 days off treatment from Day 15-21).
  Interventions: Drug: TQB2858 injection; Drug: Anlotinib Hydrochloride Capsule; Drug: Gemcitabine hydrochloride for injection; Drug: Paclitaxel for injection (albumin bound)

INTERVENTIONS:
Drug: TQB2858 injection — TQB2858 injection is a programmed cell death 1 ligand 1 (PD-L1)/transforming growth factor-β bispecific antibody.
Drug: Anlotinib Hydrochloride Capsule — Anlotinib hydrochloride is a muti-target tyrosine kinase inhibitor.
Drug: Gemcitabine hydrochloride for injection — Chemotherapy medicine for metastatic pancreatic cancer
Drug: Paclitaxel for injection (albumin bound) — Chemotherapy medicine for metastatic pancreatic cancer

SUMMARY:
This study is divided into three phases: single-dose exploration, combination dosage exploration and cohort expansion. The Single-dose exploration stage aims to evaluate the tolerability of TQB2858 injection in subjects with advanced pancreatic carcinoma. The Combination dosage exploration stage aims to evaluate the tolerance of TQB2858 injection combined with chemotherapy in patients with metastatic pancreatic cancer. The cohort expansion phase aims to evaluate the preliminary efficacy of TQB2858 injection combined with gemcitabine, albumin paclitaxel, and with or without anlotinib in patients with metastatic pancreatic cancer，and to explore treatment-related biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients voluntarily joined the study and signed the informed consent；
* 2. Aged: 18 ~ 75 years old；
* 3. Phase 1:patients who have failed to receive at least 1 line of system chemotherapy in the past or the investigator believes that they are not suitable for receiving systemic chemotherapy; The first cohort and second cohort of Phase 2 and of Phase 3: newly diagnosed patients with metastatic pancreatic cancer confirmed by tissue or cytology; The third cohort of Phase 3: patients with metastatic pancreatic cancer who have undergone first-line FOLFIRINOX or FOLFIRINOX+BRCA mutation targeted therapy or PD-1/PD-L1 treatment failure;
* 4. Confirmed to have at least one measurable lesion according to the Response Evaluation Criteria in Solid Tumours (RECIST) 1.1
* 5. Physical condition score( Eastern Cooperative Oncology Group(ECOG) score): 0~1，estimated survival time ≥ 3 months；
* 6. The main organs are functioning normally；
* 7. Women of childbearing age must be negative for serum or urine human chorionic gonadotropin (HCG) within 7 days prior to study enrollment and must be non-lactating; Patients should agree to use contraception during the study period and for 6 months after the study period；

Exclusion Criteria:

* (1) Concomitant disease and medical history:

  1. Unmitigated toxic reactions above the Common Terminology Criteria for Adverse Events (CTCAE) grade 1 due to any prior treatment, excluding hair loss and peripheral sensory nerve disorders;;
  2. Severe organ failure;
  3. Has developed other malignant tumors within 5 years or is currently suffering from the same tumor;
  4. Received major surgical treatment or significant traumatic injury (excluding needle biopsy) within 28 days prior to the commencement of study treatment;
  5. Long-term unhealed wounds or fractures;
  6. Active bleeding or researchers believe that the risk of bleeding is higher;
  7. The occurrence of arterial/venous thrombosis events within 6 months, such as cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction), deep venous thrombosis and pulmonary embolism;
  8. People with a history of psychotropic substance abuse and inability to quit or with mental disorders;
  9. Symptomatic interstitial lung disease, and conditions that may cause drug pulmonary toxicity or related pneumonia;
  10. Subjects with any severe and/or uncontrolled disease;
* (2) Tumor-related symptoms and treatment:

  1. Had undergone surgery, chemotherapy, radiation or other anticancer therapy within 4 weeks prior to the start of study treatment (washout period was calculated from the end of the last treatment);
  2. Computed tomography (CT) or Magnetic resonance imaging (MRI) shows that the tumor has invaded important blood vessels or the investigator has determined that the tumor is likely to invade important blood vessels and cause fatal hemorrhage during the follow-up study;
  3. Patients with brain metastases whose symptoms stabilized less than 4 weeks after discontinuation of dehydrants and steroids;
* (3) Research Treatment Related:

  1. Previous history of severe allergy to macromolecular drugs or known components of TQB2858 injection;
  2. Participants had participated in other antitumor drug clinical trials in the previous 4 weeks;
  3. Have been diagnosed with immunodeficiency or are receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy (dose of >10mg/ day prednisone or other equivalent efficacy hormone), and continued to use within 2 weeks of the first administration;
  4. A history of live attenuated vaccine vaccination within 28 days prior to the study treatment initiation or a planned live attenuated vaccine vaccination during the study period;
  5. Study the occurrence of active autoimmune disease requiring systemic treatment (e.g., use of palliative drugs, corticosteroids, or immunosuppressants) within 2 years prior to treatment initiation；
* (4) Participated in other anti-tumor drug clinical trials within 4 weeks before the first medication or less than 5 drug half-lives；
* (5) Subject who, in the Investigator's judgment, has a concomitant disease that seriously endangers the subject's safety or affects the completion of the study, or is considered unsuitable for inclusion for other reasons；

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-11-27 (Actual); Study Completion 2023-11-27 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | Baseline up to 3 weeks
  Grade 3 or 4 adverse events related to the study drug that occurred during cycle 1
Recommended phase II dose (RP2D) | Baseline up to 3 weeks
  Recommended dose for phase II
Overall response rate (ORR) | Baseline up to 30 weeks
  ORR refers to the percentage of complete response (CR) or partial response (PR) subjects determined by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 or iRECIST (CR and PR under iRECIST criteria can occur after imaging disease progression).

SECONDARY OUTCOMES:
Adverse event rate | Baseline up to 96 weeks
  The occurrence of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs).
Disease control rate (DCR) | Baseline up to 30 weeks
  DCR refers to the percentage of subjects with CR, PR, or stable disease (SD) of 6 weeks or more as determined by RECIST 1.1 or iRECIST (CR, PR, SD under iRECIST criteria can occur after imaging disease progression).
Duration of Response (DOR) | Baseline up to 30 weeks
  DOR will be defined as median number of months from date of first documented objective response until first documented sign of disease progression or death due to any causes.
Progression-Free Survival (PFS) | Baseline up to 30 weeks
  PFS will be defined as median number of months from the date of randomization until the first documented sign of disease progression or death due to any causes, whichever occurs first.
Overall survival (OS) | Baseline up to 96 weeks
  From randomization to the time of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China